CLINICAL TRIAL: NCT06438627
Title: Efficacy and Safety of Nab-Paclitaxel, Cisplatin, and Capecitabine Chemotherapy Combined With Apatinib and Camrelizumab vs Gemcitabine, Cisplatin Combined With Camrelizumab for Induction Chemotherapy Followed by Concurrent Chemoradiotherapy in High-Risk Nasopharyngeal Carcinoma: A Prospective, Controlled, Open-Label, Multicenter Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of TPC+Apatinib+Camrelizumab vs GP+ Camrelizumab for High-Risk Nasopharyngeal Carcinoma: A Phase 3 Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: XIANG YANQUN (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-267-02
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPC+Apatinib+Camrelizumab (Experimental): Radiation: IMRT Drug: Nab-Paclitaxel, Cisplatin, and Capecitabine Chemotherapy Combined With Apatinib and Camrelizumab (Induction chemotherapy)
  Interventions: Drug: TPC combined with Apatinib and Camrelizumab
- GP+ Camrelizumab (Active Comparator): Radiation: IMRT Drug: Gemcitabine, Cisplatin Combined With Camrelizumab (Induction chemotherapy)
  Interventions: Drug: GP Combined With Camrelizumab

INTERVENTIONS:
Drug: TPC combined with Apatinib and Camrelizumab — Nab-Paclitaxel, Cisplatin, and Capecitabine Chemotherapy Combined With Apatinib and Camrelizumab
  Arms: TPC+Apatinib+Camrelizumab
Drug: GP Combined With Camrelizumab — Gemcitabine, Cisplatin regimen Combined With Camrelizumab
  Arms: GP+ Camrelizumab

SUMMARY:
This study aims to evaluate the efficacy and safety of the TPC regimen (nab-paclitaxel, cisplatin, and capecitabine) combined with apatinib and camrelizumab versus the GP regimen (gemcitabine and cisplatin) combined with camrelizumab for the treatment of high-risk regionally advanced nasopharyngeal carcinoma with a high risk of distant metastasis. The evaluation will be conducted through a prospective, controlled, open-label, multicenter phase 3 clinical trial in areas with high incidence of nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
IMPORTANCE: Safe and effective therapies for untreated, advanced locally advanced nasopharyngeal carcinoma remain an unmet need.

OBJECTIVE:This study aims to evaluate the efficacy and safety of the TPC regimen (nab-paclitaxel, cisplatin, and capecitabine) combined with apatinib and camrelizumab versus the GP regimen (gemcitabine and cisplatin) combined with camrelizumab for the treatment of high-risk regionally advanced nasopharyngeal carcinoma with a high risk of distant metastasis. The evaluation will be conducted through a prospective, controlled, open-label, multicenter phase 3 clinical trial in areas with high incidence of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed WHO type II or III;
2. Staging TanyN3M0 (UICC/AJCC 8th edition);
3. Treatment-naive patients with no history of other malignancies;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
5. Age 18-65 years;
6. Neutrophils ≥1.5×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥90 g/L, transaminases <2.5 times the upper limit of normal, total bilirubin <1.5 times the upper limit of normal, creatinine <1.5 times the upper limit of normal; activated partial thromboplastin time and international normalized ratio <1.5 times the upper limit of normal;
7. Signed informed consent form.

Exclusion Criteria:

1. Known or suspected allergy to the study drugs, or pregnant/perinatal women;
2. Inability to comply with regular follow-up due to psychological, social, familial, or geographical reasons;
3. Severe dysfunction of critical organs such as the heart, lungs, liver, or kidneys (e.g., decompensated heart, lung, renal, or liver failure) that precludes tolerance to chemoradiotherapy;
4. Severe uncontrolled infection or internal medical disease;
5. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); untreated active hepatitis (hepatitis B defined as HBV-DNA ≥500 IU/ml, exclusion if normal liver function and on antiviral medication for more than one week; hepatitis C defined as HCV-RNA above the lower limit of detection) or coinfection with hepatitis B and C;
6. Factors affecting drug administration, distribution, metabolism, or excretion such as psychiatric disorders, central nervous system abnormalities, chronic diarrhea, ascites, or pleural effusion;
7. Poorly controlled hypertension despite antihypertensive treatment (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg);
8. Long-term use of immunosuppressants post-organ transplantation;
9. Known history of substance abuse or drug addiction;
10. History of other malignancies prior to enrollment;
11. Presence of other severe physical or mental illnesses or abnormal laboratory findings that may increase the risk of study participation, interfere with study results, or deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
3-years FFS | up to 3 years
  3-years failure-free survival rate

SECONDARY OUTCOMES:
DMFS | up to 3 years
  Distant metastasis-free survival rate
OS | up to 3 years
  Overall survival rate
LRFS | up to 3 years
  locoregional progression-free survival rate
ORR | up to 3 years
  Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Yanqun Xiang, Principal Investigator — SunYat-sen U
Locations (2):
- China (2):
  - SunYat-senU, Guangzhou, Guangdong
  - Sun Yat sen Memorial Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No